CLINICAL TRIAL: NCT02736838
Title: Peripheral Perfusion and Oxygenation in Areas of Risk of Skin Integrity Impairment Exposed to Pressure Patterns. A Phase I Trial (POTER-DIC)
Brief Title: Peripheral Perfusion and Oxygenation in Areas of Risk of Skin Integrity Impairment Exposed to Pressure Patterns.
Acronym: POTER-DIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Malaga (Other)
Collaborators: Health Service of Andalucia (Other Government)
Responsible Party: Principal Investigator, JOSE MIGUEL MORALES ASENCIO, PhD, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI15/02016
Record Dates: First submitted 2016-02-25; First posted 2016-04-13 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Pressure Ulcer
Keywords: Pressure; Pressure Ulcer; Skin perfusion; Skin oxygenation
MeSH Terms: conditions — Pressure Ulcer | interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase I (Experimental): Interventions: Different positions will be applied to subjects to measure preipheral tissue oxygenation, pressure, and changes in microvascular flow. Subjects will be placed up to 4 hours in each of the standard positions for the experiment: supine decubitus (SD) right lateral decubitus (RLD), left lateral decubitus (LLD). SD measurements will be made at 0, 30 and 45 degrees of inclination to bed. RLD and LLD positions will be evaluated with a body inclination of 30 and 90ª. The subjects will lie down on a memory foam mattress for an articulated bed, as are commonly used at home, residential or hospital care. Between the subject and the mattress will be inserted the pressure measuring surface. Measurements in each position will be made during intervals of 0-4 hours in the same position (SD-RLD-LLD) in each of the inclinations of the bed (0º, 30°, 45 °) or body (30º, 90º), respectively.
  Interventions: Device: tcpO2; Device: Laser Doppler

INTERVENTIONS:
Device: tcpO2 — Skin oxygenation will be measured by tcpO2, and microvascular flow with Laser Doppler. Measurements will be made inserting probes in sacrum, trochanters, elbows and heels, before and after the end of each decubitus lying period, and in every position and angle. Pressure: Continuous pressure measurements will be made in sacrum, trochanters, elbows and heels. Measures will be carried out at sessions separated at intervals of 7 days, with 0 to 4 hours of experimental exposure to pressure, different bed angles (0º, 30º, 45º), and lateral decubitus tilts (30, 90). Bioimpedance will be performed at baseline early in the morning, fasting and after emptying the bladder. Subjects will be lying without clothes, in a supine position on the bed, with a distance of at least 25 cm between thighs. The measurement will be made in single frequency mode (50 kHz , 400 μARMS) with a tetrapolar electrode arrangement.
Device: Laser Doppler

SUMMARY:
Objectives: 1. To analyze the changes in peripheral tissue oxygenation in tissues subjected to different pressure regimes in healthy humans. 2. To analyze changes in microvascular flow in peripheral tissues subjected to different pressure regimes in healthy humans. 3. To determine thresholds of tissue perfusion flow and transcutaneous oxygen depending on exposure levels and angling pressure in healthy volunteers. 4. To evaluate the distribution of tissue perfusion flow and transcutaneous oxygenation in real clinical situations in residential care and acute hospital care in patients at risk for impaired skin integrity.

Methodology:

Experimental non-controlled, non-randomized study in two phases: preclinical and clinical. The first phase, will be conducted in healthy volunteers and the second, in patients at risk for impaired skin integrity. Vascular flow, tissue oxygenation and local temperature in areas at risk of pressure ulcers by Doppler laser will be evaluated in subjects lying on a capacitive surface to measure pressure with 10,249 points of measurement, which will be subject to different body systems to generate different levels of pressure and monitor changes in tissue perfusion and oxygenation up to 4 hours, to know the implications for repositioning interventions in patients at risk.

DETAILED DESCRIPTION:
Sample: the preclinical phase will be conducted in 20 healthy volunteers enrolled in the Faculty of Health Sciences of the University of Malaga. Clinical phase will take place in 12 subjects admitted to acute hospitalization in 'Costa del Sol' Health Agency and 12 subjects admitted to nursing homes in the District of Primary Knowing this information will identify different thresholds start in peripheral microcirculation disorders associated with various systems of body position and consequent pressure levels. This particular seems a reasonable need from baseline parameters allow to further explore specific situations of tissue injury and isolate direct and indirect causal factors. It is also necessary to conduct the study in subjects from different environments (home, hospital) to determine under real clinical practice how these parameters behave and how it can affect common procedures performed in clinical practice, such as repositioning or using pressure surfaces. This sample of 24 subjects was calculated taking into account a change in the capillary flow of 30% between baseline and the first hour of exposure to pressure, according to data of Kallman et al. (15) with an 80% output and statistical confidence level of 95%. In total, each subject will provide a total of 28 hours of measurement.

Phase 1: Inclusion criteria:Healthy volunteers, between 20 and 65 years old, with no cardiovascular, neurological, digestive, endocrine, renal, gynecological, respiratory, hematologic, infectious, dermatological, autoimmune or diagnosed musculoskeletal disease or functional limitations, with tissue integrity and BMI between 18.5 to 25.9 kg/cm2 without scars in the sacred, back-lumbar, trochanteric, heels, elbows and shoulder blades areas.

Exclusion criteria: The usual consumption for any reason of alpha-beta-blocking agents, or alpha-beta agonists, or directly or indirectly vasodilator-vasoconstrictor action drugs of any kind, anticoagulants, topical or systemic steroids, presence of pacemakers or implantable defibrillator, smoking, high consumption of alcohol (>20g/week), presence of tattoos in the areas of measurement, and lower limb amputation

Phase 2: Inclusion criteria: Patients admitted to acute hospitalization, with risk of skin integrity deterioration assessed by Braden scale (punctuation lower than 16) without pressure ulcers, who agree to participate in the study. Exclusion criteria: presence infusion of vasoactive drugs at the time of the study (dopamine, epinephrine, norepinephrine, dobutamine, nitroprusside, nitroglycerin, calcium channel blockers, ACE inhibitors). Regular oral treatment of alpha and beta-blockers and/or agonists or calcium channel blockers, nitrates, ACE inhibitors, angiotensin, renin inhibitors, diuretics, SSRIs, NSAIDs, will be accepted. Also patients with pacemakers and/or implanted defibrillator, fever, anemia with Hb <10g/dl, hypotension with systolic blood pressure <80 mmHg, presence of transfusions in the past 4 weeks, consumption and derivatives of erythropoietin, iron supplements, oral or parenteral anticoagulants will be excluded.

Interventions: Different positions will be applied to subjects in order to measure preipheral tissue oxygenation, pressure, and changes in microvascular flow.

The subject will be placed in each of the standard positions for the experiment: supine decubitus (SD) right lateral decubitus (RLD), left lateral decubitus (LLD). SD measurements will be made at 0, 30 and 45 degrees of inclination to bed. RLD and LLD positions will be evaluated with a body inclination of 30 and 90 degrees, aided by pillows, as is done in routine clinical practice. The subjects will lie down on a memory foam mattress for an articulated bed, as are commonly used at home, residential or hospital care. Between the subject and the mattress will be inserted the pressure measuring surface. Measurements in each position will be made during intervals of 0-4 hours in the same position (SD-RLD-LLD) in each of the inclinations of the bed (0º, 30°, 45 °) or body (30º, 90º), respectively.

In case of patients, if the institutional protocol sets repositioning with a frequency of less than 4 hours, measurements will be made to the maximum that is set in each protocol. Otherwise, the maximum time for each position will be 4 hours.

Measuring instruments:

Pressure measurements will be made with the XSENSOR PX100: 64.160.02 (31.2 x 203.2 cm) pressure sensor, with 12.7 mm of space resolution of, which has 10,240 measuring points. The pressure sensor is composed with two perpendicularly oriented networks of parallel conductive strips, which are separated by a fine compressible elastomer. The intersection of two strips forms a capacitive node, determined by the surface of intersection of the two strips, and the distance separation between them, and with the elastomer. When pressure is applied to the node, the elastomer is compressed, the bands approach and capacity increases. This change in capacitance is correlated with pressure through a calibration process. The pressure range that is able to detect varies between 0.2 to 3.87 psi.

Tissue perfusion, oxygenation and temperature of the assessed area will be made with the system Periflux 5000, composed of 2 units of Laser Doppler Flowmetry (LDF): PeriFlux 5001, which includes the laser source; and PeriFlux 5002, which provides temperature and tissue oxygenation measurements. The information of both instruments will be collected and integrated into a software that allows the simultaneous measurement of all signals. Tissue oxygenation will be measured by transcutaneous oximetry (TcpO2), a noninvasive procedure that reflects the amount of oxygen diffuses into the capillaries through the epidermis. This process depends on the state of respiratory oxygenation, the oxygen carrying capacity of blood and the overall circulatory condition. Any deterioration in any of these three members, immediately affect the skin tissue perfusion, which allows to evaluate how these factors affect the PU risk. It is measured by an electrode that heats the underlying tissue to create a local hyperemia that intensifies blood perfusion and, consecuently, oxygen pressure increases. The heat dissolves the lipid structure of the keratinized layers of the epidermis, allowing the skin permeability to gas diffusion.

ELIGIBILITY:
Phase 1:

* Inclusion criteria:

  * Healthy volunteers, between 20 to 65 years old, both female and male participants are being studied
  * With no cardiovascular, neurological, digestive, endocrine, renal, gynecological, respiratory, hematologic, infectious, dermatological, autoimmune or diagnosed musculoskeletal disease or functional limitations,
  * With tissue integrity and BMI between 18.5 to 25.9 kg/cm2 without scars in the sacred, back-lumbar, trochanteric, heels, elbows and shoulder blades areas.
* Exclusion criteria:

  * The usual consumption for any reason of alpha-beta-blocking agents, or alpha-beta agonists,
  * Or directly or indirectly vasodilator-vasoconstrictor action drugs of any kind, •Anticoagulants,
  * Topical or systemic steroids,
  * Presence of pacemakers or implantable defibrillator,
  * Smoking,
  * High consumption of alcohol (>20g/week),
  * Presence of tattoos in the areas of measurement,
  * Lower limb amputation

Phase 2:

* Inclusion criteria:

  * Patients (both female and male), between 18 to 85 years old, admitted to acute hospitalization, with risk of skin integrity deterioration assessed by Braden scale (punctuation lower than 16)
  * Without pressure ulcers,
  * Who agree to participate in the study.
* Exclusion criteria:

  * Presence infusion of vasoactive drugs at the time of the study (dopamine, epinephrine, norepinephrine, dobutamine, nitroprusside, nitroglycerin, calcium channel blockers, ACE inhibitors).
  * Regular oral treatment of alpha and beta-blockers
  * And/or agonists or calcium channel blockers, Nitrates, ACE inhibitors, Angiotensin, Renin inhibitors, Diuretics, SSRIs, NSAIDs, will be accepted.
  * Also patients with pacemakers and/or implanted defibrillator,
  * Fever,
  * Anemia with Hb <10g/dl,
  * Hypotension with systolic blood pressure <80 mmHg,
  * Presence of transfusions in the past 4 weeks,
  * Consumption and derivatives of erythropoietin, iron supplements,
  * Oral or parenteral anticoagulants will be excluded.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Peripheral tissue oxygenation (transcutaneous oxygen) | Change from Baseline in each four hour session of the eleven measurement periods along days 1-2-3-4-5. From September 2016 to May 2017
  Local noninvasive measurement reflecting the amount of O2 that has diffused from the capillaries, through the epidermis to a Clark-tupe electrode at the measuring site.

SECONDARY OUTCOMES:
Microvascular flow in peripheral tissues | Change from Baseline in each four hour session of the eleven measurement periods along days 1-2-3-4-5. From September 2016 to May 2017
  Non invasive measurement through Laser Doppler, using a diode laser emitting continuous divergent radiation. The PeriFlux System 5000 equipped with PF 5010 LDPM Unit(s) is classified in USA as a class 1 laser product according to FDA CFR 1040.10. In Europe, the instrument is classified as a Class 1 laser product according to IEC 60825-1:2007. An optical fiber leads light generated by a laser to the LDPM probe tip, which rests against the tissue. The beam of light will enter the tissue and become scattered. Blood cells moving within the volume illuminated by the beam will cause the light to change frequency. This change in frequency is called a Doppler shift.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia García-Mayor, PhD, Principal Investigator — Faculty of Health Sciences, University of Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coleman S, Gorecki C, Nelson EA, Closs SJ, Defloor T, Halfens R, Farrin A, Brown J, Schoonhoven L, Nixon J. Patient risk factors for pressure ulcer development: systematic review. Int J Nurs Stud. 2013 Jul;50(7):974-1003. doi: 10.1016/j.ijnurstu.2012.11.019. Epub 2013 Feb 1. PMID 23375662
- [Background] Coleman S, Nixon J, Keen J, Wilson L, McGinnis E, Dealey C, Stubbs N, Farrin A, Dowding D, Schols JM, Cuddigan J, Berlowitz D, Jude E, Vowden P, Schoonhoven L, Bader DL, Gefen A, Oomens CW, Nelson EA. A new pressure ulcer conceptual framework. J Adv Nurs. 2014 Oct;70(10):2222-34. doi: 10.1111/jan.12405. Epub 2014 Mar 31. PMID 24684197
- [Background] Stekelenburg A, Strijkers GJ, Parusel H, Bader DL, Nicolay K, Oomens CW. Role of ischemia and deformation in the onset of compression-induced deep tissue injury: MRI-based studies in a rat model. J Appl Physiol (1985). 2007 May;102(5):2002-11. doi: 10.1152/japplphysiol.01115.2006. Epub 2007 Jan 25. PMID 17255369
- [Background] Moore ZE, Cowman S. Repositioning for treating pressure ulcers. Cochrane Database Syst Rev. 2015 Jan 5;1(1):CD006898. doi: 10.1002/14651858.CD006898.pub4. PMID 25561248
- [Background] Gillespie BM, Chaboyer WP, McInnes E, Kent B, Whitty JA, Thalib L. Repositioning for pressure ulcer prevention in adults. Cochrane Database Syst Rev. 2014 Apr 3;2014(4):CD009958. doi: 10.1002/14651858.CD009958.pub2. PMID 24700291
- [Background] Chou R, Dana T, Bougatsos C, Blazina I, Starmer AJ, Reitel K, Buckley DI. Pressure ulcer risk assessment and prevention: a systematic comparative effectiveness review. Ann Intern Med. 2013 Jul 2;159(1):28-38. doi: 10.7326/0003-4819-159-1-201307020-00006. PMID 23817702
- [Background] Nakagami G, Sanada H, Iizaka S, Kadono T, Higashino T, Koyanagi H, Haga N. Predicting delayed pressure ulcer healing using thermography: a prospective cohort study. J Wound Care. 2010 Nov;19(11):465-6, 468, 470 passim. doi: 10.12968/jowc.2010.19.11.79695. PMID 21135794
- [Background] Farid KJ, Winkelman C, Rizkala A, Jones K. Using temperature of pressure-related intact discolored areas of skin to detect deep tissue injury: an observational, retrospective, correlational study. Ostomy Wound Manage. 2012 Aug;58(8):20-31. PMID 22879313
- [Background] Kokate JY, Leland KJ, Held AM, Hansen GL, Kveen GL, Johnson BA, Wilke MS, Sparrow EM, Iaizzo PA. Temperature-modulated pressure ulcers: a porcine model. Arch Phys Med Rehabil. 1995 Jul;76(7):666-73. doi: 10.1016/s0003-9993(95)80637-7. PMID 7605187
- [Background] Behrendt R, Ghaznavi AM, Mahan M, Craft S, Siddiqui A. Continuous bedside pressure mapping and rates of hospital-associated pressure ulcers in a medical intensive care unit. Am J Crit Care. 2014 Mar;23(2):127-33. doi: 10.4037/ajcc2014192. PMID 24585161
- [Background] Swisher SL, Lin MC, Liao A, Leeflang EJ, Khan Y, Pavinatto FJ, Mann K, Naujokas A, Young D, Roy S, Harrison MR, Arias AC, Subramanian V, Maharbiz MM. Impedance sensing device enables early detection of pressure ulcers in vivo. Nat Commun. 2015 Mar 17;6:6575. doi: 10.1038/ncomms7575. PMID 25779688
- [Background] Sarnik S, Hofirek I, Sochor O. Laser Doppler fluxmetry. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2007 Jun;151(1):143-6. doi: 10.5507/bp.2007.028. PMID 17690759
- [Background] Kallman U, Engstrom M, Bergstrand S, Ek AC, Fredrikson M, Lindberg LG, Lindgren M. The effects of different lying positions on interface pressure, skin temperature, and tissue blood flow in nursing home residents. Biol Res Nurs. 2015 Mar;17(2):142-51. doi: 10.1177/1099800414540515. Epub 2014 Jul 18. PMID 25037449
- [Derived] Gomez-Gonzalez AJ, Morilla-Herrera JC, Lupianez-Perez I, Morales-Asencio JM, Garcia-Mayor S, Leon-Campos A, Marfil-Gomez R, Aranda-Gallardo M, Moya-Suarez AB, Kaknani-Uttumchandani S. Perfusion, tissue oxygenation and peripheral temperature in the skin of heels of healthy participants exposed to pressure: a quasi-experimental study. J Adv Nurs. 2020 Feb;76(2):654-663. doi: 10.1111/jan.14250. Epub 2019 Nov 20. PMID 31651050
- [Derived] Garcia-Mayor S, Morilla-Herrera JC, Lupianez-Perez I, Kaknani Uttumchandani S, Leon Campos A, Aranda-Gallardo M, Moya-Suarez AB, Morales-Asencio JM. Peripheral perfusion and oxygenation in areas of risk of skin integrity impairment exposed to pressure patterns. A phase I trial (POTER Study). J Adv Nurs. 2018 Feb;74(2):465-471. doi: 10.1111/jan.13414. Epub 2017 Sep 15. PMID 28792613